CLINICAL TRIAL: NCT07079384
Title: Evaluation of Patient Comfort and Satisfaction After the Construction of Maxillary Obturator Prosthesis for Limited Mouth Opening in Maxillofacial Cases With Different Approaches: Cross Over Randomized Clinical Trial
Brief Title: Evaluation of Patient Satisfaction After the Construction of Maxillary Obturator Prosthesis for Limited Mouth Opening in Maxillofacial Cases : Cross Over Randomized Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: R.25.04.3
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Patient Satisfaction; Maxilofacial
Keywords: maxillofacial cases; limited mouth opening; obturator
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients will receive obturator fabricated by the conventional method (Active Comparator): Hollow bulb obturator plate (using lost salt technique) will be made over the obtained cast. The obturator will be finished & polished, and delivered to the patient.
  Interventions: Other: The patient will be instructed about wearing the prosthesis. First, seat the prosthesis in a posterior undercut, then rotate the prosthesis slightly superiorly in the defect area and engage the anteri
- patients will receive obturator fabricated by the digital method (Active Comparator): Extraoral scanning will be done for the cast and the virtual model will be generated by using the digital software and exported as a standard tessellation language (STL) file. The STL file was imported into CAD software
  - The designed two parts will be exported as an STL file and upload into the 3D printer software.
  Interventions: Other: The patient will be instructed about wearing the prosthesis. First, seat the prosthesis in a posterior undercut, then rotate the prosthesis slightly superiorly in the defect area and engage the anteri

INTERVENTIONS:
Other: The patient will be instructed about wearing the prosthesis. First, seat the prosthesis in a posterior undercut, then rotate the prosthesis slightly superiorly in the defect area and engage the anteri — * The obturator will then be printed using Denture Base Resin and teeth.
  * The printed obturator will be tried in, two magnets, one anteriorly and another posteriorly will be picked up then inserted into the patient mouth.
  * The patient will be again instructed regarding the care of the prosthesis and hygiene maintenance as formerly. The patient will also be instructed to wear the obturator plate first, and once this is comfortably seated, the denture part will be inserted. During removal, the patient will be instructed to first remove the denture part gently to disengage the magnetic attraction after the obturator part as formerly instructed. The patient will be recalle

SUMMARY:
A patient's quality of life is frequently negatively impacted by oral cancer, which is a serious condition. Treatment for oral cancer, which includes radiation, chemotherapy, and surgery, can result in several oral complications. The risk of impression material becoming lodged in undercuts and the challenges in retrieving the material would be inconvenient for both the patient and the dentist. Therefore, a digital pathway was chosen for the prosthesis fabrication process So, the present study aims to investigate the patient comfort and satisfaction after the construction of maxillary interim obturator for radiation-induced trismus in maxillofacial cases with different approaches: conventional and digital fabrication processes.

DETAILED DESCRIPTION:
A patient's quality of life is frequently negatively impacted by oral cancer, which is a serious condition. Treatment for oral cancer, which includes radiation, chemotherapy, and surgery, can result in several oral complications, including trismus, xerostomia, dysgeusia, odontogenic infections, and osteoradionecrosis.

Aim: the present study aims to investigate the patient comfort and satisfaction after the construction of maxillary interim obturator for radiation-induced trismus in maxillofacial cases with different approaches: conventional and digital fabrication processes.

Methodology: The present crossover study will be conducted on 30 maxillofacial patients with maxillary defect with limited mouth opening, aged between 50 -65 years, will be selected for the study from the Maxillofacial clinic of the Prosthodontic Department, Faculty of Dentistry, Mansoura University.A preliminary impression of the maxillary defect will be made with a high-viscosity irreversible hydrocolloid, covering all the margins of the defect and blocking all unfavorable undercuts with wet gauge piece.In a simple randomized method, 15 patients will receive obturator fabricated by the digital method.The other 15 patients will receive obturator fabricated by the conventional method Patient comfort and satisfaction by visual analogue scale (VAS), and Gothenburg Trismus Questionnaire (GTQ) at follow-up periods as follows: T0 immediately after insertion of obturator, T1= three months after insertion of obturator, T2=six months after insertion of obturator.

ELIGIBILITY:
Inclusion Criteria:

Patient with unilateral total maxillectomy.

Free from any signs of inflammation in the defect area. The defect size is large.

Exclusion Criteria:

Patient is still receiving radiation. The defect size is small. Defects result from trauma.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-10-12 (Estimated); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
VAS of pain | six months
  1-The patients used a visual analogue scale (VAS) to self-assess their level of pain, with 10 representing the most severe pain.

SECONDARY OUTCOMES:
Gothenburg Trismus Questionnaire (GTQ) | six months
  The GTQ seems to be the most reliable tool for measuring trismus that is now available since a more comprehensive assessment of trismus and its treatment effects requires a multidimensional, self-administered, trismus-specific measure, which is what the GTQ offers. Its wider applicability would allow for consistent recording of trismus-related issues and a chance to get patient feedback on treatment results. The updated GTQ version had 13 items spread over three domains: eating restriction (4 items), jaw-related issues (6 items), and muscular stress (3 items). Scores on the calculated scale vary from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Ahmed Aboelez, Assistant professor, Principal Investigator — Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboelez MA, Ibrahim AM, ElSawy MA, Sayed El-Khamisy NE. Efficiency of different treatment modalities on radiation induced trismus for maxillofacial cases: a parallel randomized clinical trial. BMC Oral Health. 2025 Mar 4;25(1):332. doi: 10.1186/s12903-025-05600-7. PMID 40038715